CLINICAL TRIAL: NCT07290816
Title: Effect of Non-invasive Neuromodulation on the Quality of Bowel Cleansing: a Randomized, Controlled, Double-blind Clinical Study
Brief Title: Effect of Non-invasive Neuromodulation on the Quality of Intestinal Cleansing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023YS-077 Amendment 1
Record Dates: First submitted 2025-05-29; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-05

CONDITIONS: Intestinal Polyps
Keywords: Bowel Preparation; Noninvasive electrical neuromodulation
MeSH Terms: conditions — Intestinal Polyps

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trial Group 1 (Experimental): Bowel pacing (specific location and parameters) and ST36 acupoint stimulation (specific location and intensity) were used the day before the examination; 2L of PEG was taken the night before the examination and on the day of the examination, and 30 ml of simethicone was taken orally immediately after all of the 4L of PEG had been taken. Colonoscopy was completed within 2-6 hours after bowel preparation was completed.
  Interventions: Other: Intestinal pacing + ST36 acupoint stimulation
- Trial Group 2 (Experimental): Sham acupoint bowel pacing and sham ST36 acupoint stimulation were used the day before the examination (electrode pads were offset and current switch was not turned on; 2L of PEG was taken the night before and on the day of the examination, respectively, and 30 ml of simethicone was taken orally immediately after all of the 4L of PEG had been taken. Colonoscopy was completed within 2-6 hours after bowel preparation was completed.
  Interventions: Other: Sham acupoint intestinal pacing + sham ST36 acupoint stimulation
- Control Group (No Intervention): Only conventional treatment was used, with 2 portions of 2000 ml PEG taken with fasting starting at 19:00 pm the night before the examination and required to be taken within 2 hours. On the day of the examination, 2 doses of 2000 ml of PEG were taken orally starting 3-5 hours before the colonoscopy procedure, which was required to be completed within 2 hours, and 30 ml of simethicone was taken orally as soon as the subject had finished taking the laxative, and all bowel preparations had to be completed more than 2 hours and less than 6 hours before the colonoscopy procedure, and if the time limit was exceeded the subject was excluded from the study.

INTERVENTIONS:
Other: Intestinal pacing + ST36 acupoint stimulation — The day before the examination began a real stimulation treatment, namely, intestinal pacing (① location: positive pole placed on the navel (the line between the raphe and navel) 1 to 2 cm, the negative pole in the raphe and the navel line at the midpoint of the right 4 to 10 cm; ② parameters: the intestinal frequency: 2.4-3.7 cpm, the first time the frequency of use of 3.0 cpm, treatment of the base wave intensity of 0-15 gears, the first time to use the intestinal treatment intensity of 10 gears) , acupoint stimulation (① location: treatment sheet attached to both legs ST36 acupoints, i.e., four transverse fingers below the eye of the outer knee, 4 transverse fingers next to the tibia; ② parameters: the first use of acupoint intensity 30%, to the patient's self-conscious stimulation points have a slight pinprick sensation, lifting sensation, warm sensation is appropriate).
  Arms: Trial Group 1
Other: Sham acupoint intestinal pacing + sham ST36 acupoint stimulation — A sham stimulation treatment was started one day before the examination, i.e., intestinal pacing treatment with the electrode pads offset to the lumbar side to stimulate the sham acupoints, and acupoint stimulation with the treatment pads applied to the ST36 acupoints but without turning on the current switch.
  Arms: Trial Group 2

SUMMARY:
To clarify whether non-invasive neuromodulation for assisted bowel preparation can improve the quality of bowel preparation, to explore the possible mechanisms by which TEA improves the quality of bowel preparation, and to assess its safety, as well as subjects' tolerance, compliance and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 78 years of age, male or female;
* Intended to undergo diagnostic, screening, or surveillance colonoscopy;
* Signed written informed consent.

Exclusion Criteria:

* Severe cardiac, cerebral, pulmonary, or renal complications or a history of acute cardiac infarction within six months;
* High risk factors for bowel preparation such as history of colon surgery, BMI ≥ 28, inflammatory bowel disease, constipation (less than 3 bowel movements in the last week, and with straining to defecate, with hard stools and small amount of stools) or bowel obstruction;
* High suspicion of colorectal cancer by auxiliary examination or early warning signs and symptoms of colorectal cancer: blood in stool, black stool, unexplained anemia, significant weight loss, abdominal mass and positive rectal fingerprinting;
* The presence of surgical incisions or scars in the area where the electrostimulation treatment tablets are pasted, or near the ST36 acupoints on both legs;
* Are participating in other clinical observation trials or have participated in other clinical trials within 30 days.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-03-21 (Estimated); Study Completion 2028-03-21 (Estimated)

PRIMARY OUTCOMES:
Bowel Preparedness Score | Day 2
  Using the Boston Bowel Preparation Scale(BBPS)

SECONDARY OUTCOMES:
Polyp detection rate | Day 2
Adenoma detection rate | Day 2
Adverse reactions | Baseline and Day 2
  collected using a questionnaire
Complete Blood Count | Baseline and Day 2
C-Reactive Protein | Baseline and Day 2
Inflammatory Cytokines(TNF-α，IL-6，IL-10……) | Baseline and Day 2
Gastrointestinal Hormones (Pancreatic Polypeptide, Motilin, Vasoactive Intestinal Peptide……) | Baseline and Day 2

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No